CLINICAL TRIAL: NCT05569070
Title: Evaluation of Young United Parents
Acronym: YUP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 90AP2692-01-00
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Teen Pregnancy Prevention
Keywords: Teen Pregnancy Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided Young United Parents! (YUP!) Website Intervention (Experimental): The Guided YUP! website intervention is the treatment condition, which will involve two months of directed use of the YUP! website.
  Interventions: Other: Guided Young United Parents! Website Intervention
- Nutrition Website (Sham Comparator): The nutrition website is the control condition.
  Interventions: Other: Nutrition Website

INTERVENTIONS:
Other: Guided Young United Parents! Website Intervention — Participants assigned to Guided YUP! will receive two months of structured use of the YUP! website intervention, which involves weekly review of written and video content, meetings with near-peer mentors, use of the goal tool, interaction with the online community, and receipt of tips and affirmations.
  Arms: Guided Young United Parents! (YUP!) Website Intervention
Other: Nutrition Website — Participants assigned to the Nutrition Website will be provided with the link to the MyPlate website, which is maintained by the U.S. Department of Agriculture. At the enrollment session, participants will be given brief instruction during the enrollment session about features available on the website that may be interesting to them and encouraged to engage in any of the website or app features at whatever level they are comfortable with. No further direction will be provided to them after the enrollment session.
  Arms: Nutrition Website

SUMMARY:
The purpose of the study is to determine the impact of the offer to participate in the Young United Parents! (YUP!) intervention relative to the control condition on use of effective non-barrier contraception and frequency of vaginal sex without condoms three months after the intervention period has concluded.

DETAILED DESCRIPTION:
The Policy & Research Group (PRG) will be rigorously evaluating an innovative intervention, Young United Parents! (YUP!), which is a website-based program designed to help young parents ages 15-22 avoid unplanned, repeat pregnancy and sexually transmitted infections (STIs), reach their personal goals, and thrive in all areas of life. The mobile-optimized website contains 50 articles and over 100 personal narrative videos of highly diverse young parents and experts. The YUP! intervention includes: 1) video and written content on six topics (sexual health and birth control; healthy relationships; self-care; reaching your goals; parenting; and pregnancy and birth); 2) access to near-peer mentors; 3) a goal-setting tool; 4) daily tips, reminders, and motivational messages; 5) links and referrals to support services; and 6) membership in the YUP! online community of young parents.

PRG will conduct an implementation evaluation and an impact evaluation of a structured version of YUP!, called Guided YUP!. Guided YUP! involves a two-month program experience during which participants are directed through a dashboard on the website to review between 15-35 minutes of particular website content each week. Participants will also be paired with a near-peer mentor who will schedule virtual interactions with them every two weeks, for a total of at least five interactions over the course of the two-month intervention period. All interactions will be held via the YUP! participant dashboard and are expected to last between 5-10 minutes. The aim of these interactions is for the near-peer mentor to offer support and guidance, using motivational interviewing techniques, as the participants go through the Guided YUP! program. Additionally, Guided YUP! participants will be asked to outline and complete at least one goal during the two-month intervention period, using the goal tool on the website. Guided YUP! participants will also receive automatically generated tips and affirmations through the website and have access to the YUP! online community to participate in, if desired.

PRG will assess the efficacy of Guided YUP! using a randomized controlled trial. The study will target young mothers ages 15-20 who are currently caring for their child(ren) and not pregnant or trying to become pregnant. The primary aim of the study will be to investigate the impact of the intervention on two self-reported sexual behaviors: 1) use of effective non-barrier contraception and 2) frequency of vaginal sex without condoms. In addition, the study will include exploratory investigations of the following self-reported sexual behaviors and theoretically relevant antecedents to these behaviors: 1) frequency of sexually transmitted infection (STI) testing; 2) frequency of completely unprotected vaginal sex; 3) incidence of pregnancy; 4) incidence of STIs; 5) condom, contraceptive, and STI knowledge; 6) condom negotiation, contraceptive use, and STI testing self-efficacy; 7) condom and contraceptive use outcome expectations; and 8) perceived pregnancy fatalism. Finally, the study will explore the impact of the intervention on measures that assess participants' perceptions of their healthy relationships, self-care and well-being, goal achievement, and parenting competence.

Outcomes will be assessed using self-reported, participant-level data gathered using a structured questionnaire administered at four time points: baseline (enrollment); post-intervention (two months after baseline); three months post-intervention (five months after the baseline); and twelve months post-intervention (fourteen months after the baseline).

Starting in October 2022 and continuing for 21 months, 1400 participants from around the United States will be enrolled virtually. The final two years of the grant will be used to collect follow-up data from study participants; conduct implementation and impact evaluation analysis, reporting, and dissemination efforts.

ELIGIBILITY:
Inclusion Criteria:

* Biological female aged 15-20
* Has given birth to a child they currently provide care for
* Reports having penile-vaginal sex at least one time in past three months
* Fluent in English (able to read and comprehend the online intervention materials, which are available only in English)
* Owns or has regular access to a personal device (smartphone, laptop, tablet) with internet access
* United States resident
* Provides informed assent or consent for study participation

Exclusion Criteria:

* Currently pregnant
* Currently trying to become pregnant
* Previously registered to use the YUP! website
* Enrolled in an ongoing PRG-run TPP study
* Identified as fraudulent

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1400 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Use of effective non-barrier contraception | Assessed three months after the intervention period has ended
  Participant self-report on whether (or not) they are currently using effective non-barrier contraception (IUD, implant, oral contraceptive pill, injection, patch, or ring)
Times having vaginal sex without a condom | Assessed three months after the intervention period has ended
  Participant self-report on the number of times having vaginal sex without using a condom during the past three months

SECONDARY OUTCOMES:
Contraceptive knowledge | Assessed immediately post-intervention and three months after the intervention period has ended
  Proportion of items related to contraceptive knowledge to which the participant answers correctly
Condom knowledge | Assessed immediately post-intervention and three months after the intervention period has ended
  Proportion of items related to condom knowledge to which the participant answers correctly
STI knowledge | Assessed immediately post-intervention and three months after the intervention period has ended
  Proportion of items related to STI knowledge to which the participant answers correctly
Condom negotiation self-efficacy | Assessed immediately post-intervention and three months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of confidence in being able to negotiate condom use, with scores ranging from 1 (indicating low confidence) to 7 (indicating high confidence)
Contraceptive use self-efficacy | Assessed immediately post-intervention and three months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of confidence in being able to use contraceptives, with scores ranging from 1 (indicating low confidence) to 7 (indicating high confidence)
STI testing self-efficacy | Assessed immediately post-intervention and three months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of confidence in being able to get STI testing, with scores ranging from 1 (indicating low confidence) to 7 (indicating high confidence)
Self-care self-efficacy | Assessed immediately post-intervention and three months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of confidence in being able to take care of themselves, with scores ranging from 1 (indicating low confidence) to 7 (indicating high confidence)
Goal setting self-efficacy | Assessed immediately post-intervention and three months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of confidence in being able to set personal goals, with scores ranging from 1 (indicating low confidence) to 7 (indicating high confidence)
Condom use outcome expectations | Assessed immediately post-intervention and three months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of agreement with statements about the outcomes expected with condom use, with scores ranging from 1 (indicating low agreement) to 7 (indicating high agreement)
Contraceptive use outcome expectations | Assessed immediately post-intervention and three months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of agreement with statements about the outcomes expected with contraceptive use, with scores ranging from 1 (indicating low agreement) to 7 (indicating high agreement)
Perceived pregnancy fatalism | Assessed immediately post-intervention and three months after the intervention period has ended
  Mean score to one item that asks an individual to self-report their level of agreement with a statement related to what degree they have control over becoming pregnant, with scores ranging from 1 (indicating low agreement) to 7 (indicating high agreement)
Use of effective non-barrier contraception | Assessed twelve months after the intervention period has ended
  Participant self-report on whether (or not) they are currently using effective non-barrier contraception (IUD, implant, oral contraceptive pill, injection, patch, or ring)
Consistent use of effective non-barrier contraception | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) they have been using effective non-barrier contraception consistently for the past three months
Frequency of emergency contraception use | Assessed three and twelve months after the intervention period has ended
  Participant self-report on the number of times they have used emergency contraception after vaginal sex in the past three months
Use of effective non-barrier contraception during last vaginal sex | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) they used effective non-barrier contraception during the last time they had vaginal sex
Times having vaginal sex without a condom | Assessed twelve months after the intervention period has ended
  Participant self-report on the number of times having vaginal sex without using a condom during the past three months
Use of condoms during last vaginal sex | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) they used condoms during the last time they had vaginal sex
Times having completely unprotected during last vaginal sex | Assessed three and twelve months after the intervention period has ended
  Participant self-report on the number of times having vaginal sex with neither a condom nor effective non-barrier contraception during the past three months
Completely unprotected during last vaginal sex | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) their last vaginal sex act was completely unprotected (using neither a condom nor effective non-barrier contraception)
Dual methods of protection during recent vaginal sex | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) they used dual methods of protection (both condoms and effective non-barrier contraception) during recent vaginal sex
Dual methods of protection during last vaginal sex | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) they used dual methods of protection (both condoms and effective non-barrier contraception) during the last time they had vaginal sex
Recent STI testing | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) they received recent STI testing
Recent STI acquisition | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) they recently tested positive for STIs
Recent repeat pregnancy | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) they have been pregnant in the recent past
Recent repeat unintended pregnancy | Assessed three and twelve months after the intervention period has ended
  Participant self-report on whether (or not) they have been pregnant in the recent past with a pregnancy that was unintended
Parenting competence | Assessed immediately post-intervention and three and twelve months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of agreement with statements about their perceived competence in their ability to take care of their child(ren), with scores ranging from 1 (indicating low agreement) to 7 (indicating high agreement)
Stigma | Assessed immediately post-intervention and three and twelve months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of agreement with statements about the perceived stigma they experience due to being a young parent, with scores ranging from 1 (indicating low agreement) to 7 (indicating high agreement)
Social support | Assessed immediately post-intervention and three and twelve months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of agreement with statements about their perceived social support, with scores ranging from 1 (indicating low agreement) to 7 (indicating high agreement)
Well-being | Assessed immediately post-intervention and three and twelve months after the intervention period has ended
  Mean scale score of items that ask an individual to self-report their level of agreement with statements about their perceived well-being, with scores ranging from 1 (indicating low agreement) to 7 (indicating high agreement)
Goal attainment | Assessed immediately post-intervention and three and twelve months after the intervention period has ended
  Mean scale score of items that ask an individual to what extent statements about their ability to set and achieve goals are similar to them, with scores ranging from 1 (indicating not at all like them) to 5 (indicating exactly like them)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jenner, PhD, Principal Investigator — The Policy & Research Group
Locations (1):
- The Policy & Research Group, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes de-identified individual-level data on all study participants who contributed self-report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program components were completed). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Supporting Information: SAP
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.